CLINICAL TRIAL: NCT02236728
Title: Observational Study in Parkinson's Disease of the Primary Care Population of Patients Treated With Pramipexole by Neurologists in France (ETAP)
Brief Title: Observational Study in Parkinson's Disease of the Primary Care Population of Patients Treated With Pramipexole
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.648
Record Dates: First submitted 2014-09-10; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Parkinson's disease patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: (Sifrol®)

SUMMARY:
The primary objective of this study was to describe neurologists' population of patients treated with pramipexole and suffering from Parkinson's disease (so called 'primary care' population).

The secondary objectives were:

* Evaluate the mean dose of pramipexole prescribed under actual conditions of use depending on the severity of the disease.
* Evaluate the reasons for choosing pramipexole as treatment.
* Identify the patient profiles determining the choice of dose of pramipexole prescribed

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from idiopathic Parkinson's Disease and treated with pramipexole for at least two months, examined in consultation

Exclusion Criteria:

* Patient refusing to take part
* Patient taking part in a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neurologists' population of patients treated with pramipexole and suffering from Parkinson's disease (so called 'primary care' population)
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Patient's demographic characteristics | 9 months
Assessment of Parkinson's disease characteristics | 9 months

SECONDARY OUTCOMES:
Assessment of Severity of the Parkinson Disease (PD) | 9 months
  (levels of severity of the disease were defined with the scientific committee in 5 stages: treatment initiation phase, honeymoon phase, therapeutic insufficiency phase, start of motor complications phase and advanced motor complications phase)
Assessment of Disease Stage Stage according to Hoehn and Yahr and Unified Parkinson Disease Rating Scale III (UPDRS III) scores | 9 months
Description of the actual treatments of PD | 9 months
Evaluation for reasons for choosing pramipexole as treatment | 9 months
Assessment of Treatment history | 9 months
  3 subgroups: Initiation: no antiparkinson treatment before the implementation of pramipexole Switch: at least one dopamine agonist replaced by pramipexole Add on: pramipexole is implemented in addition to the previous treatment
Evaluation of the state of health perceived by the patient using the questionnaire EQ-5D | 9 months
Number of patients with adverse events | 9 months